CLINICAL TRIAL: NCT02504008
Title: CREATE-1 Study: CRPS Treatment Evaluation 1 Study. A Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of AXS-02 (Oral Zoledronate) Administered Orally to Subjects With Complex Regional Pain Syndrome Type I (CRPS-I)
Brief Title: CREATE-1: A Study to Assess the Efficacy and Safety of AXS-02 in Patients With CRPS-1
Acronym: CREATE-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS02-301
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Complex Regional Pain Syndrome; Reflex Sympathetic Dystrophy
Keywords: bisphosphonate; CRPS; RSD; non-opioid; CRPS-1; acute on chronic pain; chronic pain; zoledronic acid
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Chronic Pain | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXS-02 (oral zoledronate) (Experimental): Administered orally in the morning on Days 1, 8, 15, 22, 29, and 36
  Interventions: Drug: AXS-02 (oral zoledronate)
- Placebo (Placebo Comparator): Administered orally in the morning on Day 1, 8, 15, 22, 29, and 36
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-02 (oral zoledronate) — Once weekly for 6 weeks
  Arms: AXS-02 (oral zoledronate)
Drug: Placebo — Once weekly for 6 weeks
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 24-week study to evaluate the efficacy and safety of AXS-02 in patients with CRPS-I.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female of at least 18 years of age
* Recently confirmed diagnosis of CRPS-1 (Budapest criteria)
* Average pain intensity score of ≥ 5 (based on an 11-point scale [0 - 10])
* Willing and able to provide written informed consent

Key Exclusion Criteria:

* Received chronic opioid therapy within 4 weeks
* Received a sympathetic nerve block within 3 weeks
* Active litigation or a pending workers' compensation decision
* Any other clinically significant medical or pain condition (eg, Parkinson's disease, cognitive impairment, or fibromyalgia) or clinical laboratory abnormality that would in the investigator's judgment interfere with the subject's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported pain intensity | Baseline to Week 12
  Patient reported pain intensity is recorded as an average daily pain intensity using an 11-point scale (0 = no pain to 10 = worst pain possible).

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) Pain Score | Baseline to Week 12
  The BPI is a nine-question survey completed by the patient that assesses quality of life and health status. BPI scores range from 0 to 10, with higher values indicating greater pain.
Patients' Global Impression of Change (PGI-C) | Baseline to Week 12
  The PGI-C is a patient/patient's caregiver rated scale to assess the patients overall treatment response. PGI-C is a 7-point (1-7) scale rated as; very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Clinicians' Global Impression of Change (CGI-C) | Baseline to Week 12
  The CGI-C is an investigator-rated scale to assess the overall treatment response. CGI-C is a 7-point (1-7) scale rated as; very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Change in EuroQOL 5-dimensions questionnaire (EQ-5D) | Baseline to Week 12
  The EQ-5D descriptive system comprised the following 5 dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated by the patient at one of 5 levels, with level 1 indicating the best health state (no problems) and level 5 indicating worst health state (e.g., unable to walk about).
Change in Short-Form McGill Pain Questionnaire (SF-MPQ-2) | Baseline to Week 12
  The SF-MPQ-2 measures both neuropathic and nonneuropathic pain. It contains a total of 22 descriptors, which are rated on an intensity scale of 0 = None, to 10 = Worst Possible.
Change in bone turnover markers | Baseline to Week 52
  Bone turnover is measured from 2 biomarkers collected from peripheral blood samples: serum carboxy terminal telopeptide of collagen type I (CTX) and serum procollagen type I N terminal propeptide (s-P1NP).

CONTACTS AND LOCATIONS:
Locations (44):
- United States (29):
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Encinitas, California
  - La Jolla, California
  - Los Angeles, California
  - Napa, California
  - Temecula, California
  - Denver, Colorado
  - Clermont, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Canton, Georgia
  - Marietta, Georgia
  - St. Marys, Georgia
  - Meridian, Idaho
  - Chicago, Illinois
  - Louisville, Kentucky
  - Albuquerque, New Mexico
  - New York, New York
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Dallas, Texas
  - San Antonio, Texas
  - Bellevue, Washington
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (6):
  - Broadmeadow, New South Wales
  - Hurstville, New South Wales
  - Noosa, Queensland
  - Welland, South Australia
  - Clayton, Victoria
  - Nedlands, Western Australia
- Sherbrooke, Quebec, Canada
- United Kingdom (8):
  - Warrington, Cheshire
  - Darlington, County Durham
  - Lambeth, London
  - Liverpool, Merseyside
  - Norwich, Norfolk
  - Newcastle upon Tyne, Tyne and Wear
  - Glasgow
  - London